CLINICAL TRIAL: NCT07280247
Title: Acute Pulmonary Embolism Treatment With the AlphaVac Multipurpose Mechanical Aspiration System and the AlphaReturn Blood Management System: Evaluation of Safety and Effectiveness (APEX-Return)
Brief Title: Acute Pulmonary Embolism Treatment With the AlphaVac Multipurpose Mechanical Aspiration System and the AlphaReturn Blood Management System: Evaluation of Safety and Effectiveness
Acronym: APEX-Return
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-CAR-03
Record Dates: First submitted 2025-11-25; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Embolism Acute
Keywords: pulmonary embolism; alphareturn
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AlphaVac MMA F1885 System and AlphaReturn Blood Management System (Experimental): Following mechanical thrombectomy using the AlphaVac MMA System, the treating physician will filter the aspirated blood using the AlphaReturn Blood Management System and reinfuse the filtered autologous blood back into the patient.
  Interventions: Device: AlphaReturn Blood Management System

INTERVENTIONS:
Device: AlphaReturn Blood Management System — The AlphaReturn Blood Management System allows for autologous injection of aspirated blood from an AlphaVac MMA System thrombectomy procedure.

SUMMARY:
The investigation is intended to evaluate the safety and effectiveness of the AlphaReturn Blood Management System when used in conjunction with the cleared AlphaVac MMA F1885 System for the treatment of acute pulmonary embolism.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm investigational device study evaluating safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

A potential subject will be included in the study if he/she meets all the following inclusion criteria:

1. Provision of signed and dated informed consent form.
2. Subject is 18 years of age and older.
3. Subject presents clinical signs and symptoms consistent with acute intermediate-risk pulmonary embolism for less than or equal to 14 days.
4. Subject has a diagnosis of pulmonary embolism detected from computed tomography angiography (CTA).
5. Subject has a RV/LV ratio of 0.9 or higher.
6. Subject has a systolic blood pressure (SBP) of 90mmHg or higher.
7. Subject has a heart rate of 130 beats per minute (BPM) or less prior to the procedure.
8. Subject is deemed medically eligible for interventional procedure(s) per institutional guidelines and/or clinical judgment.

Exclusion Criteria:

A potential subject will be excluded from the study if he/she meets any of the following exclusion criteria:

1. Subjects who are or may be pregnant as determined by a positive pregnancy test or who are breastfeeding.
2. Subjects who have any contraindication to systemic or therapeutic doses of heparin or anticoagulants.
3. Subjects who have used thrombolytics in the 30 days prior to the baseline CTA.
4. Subjects who have pulmonary hypertension with peak pulmonary artery pressure (PAP) > 70 mmHg.
5. Subjects who have FiO2 requirement > 44% or > 6 LPM to keep oxygen saturations > 90%.
6. Subjects with hematocrit < 28% within 6 hours of index procedure.
7. Subjects with platelets count < 100,000/μL.
8. Subjects with serum creatinine > 1.8 mg/dL.
9. Subjects with International Normalized Ratio (INR) > 3.
10. Subjects who have undergone a major trauma within the past 14 days of the index procedure and have Injury Severity Score (ISS) > 15.
11. Subjects with the presence of cancer requiring active chemotherapy.
12. Subjects with known bleeding diathesis or coagulation disorder.
13. Subjects who have had a cardiovascular or pulmonary surgery within the past 7 days of index procedure.
14. Subjects with a history of severe or chronic pulmonary hypertension, uncompensated heart failure, chest irradiation, underlying lung disease that is oxygen dependent, heparin-induced thrombocytopenia (HIT) and/or chronic left heart disease with left ventricular ejection fraction ≤ 30%.
15. Subjects with known anaphylactic reaction to radiographic contrast agents that cannot be pretreated.
16. Subject requires vasopressor after fluids to keep pressure ≥ 90mmHg.
17. Subjects with left bundle branch block.
18. Subjects who have intracardiac lead in the right ventricle or atrium.
19. Evidence such as imaging or other that suggest the subject is not appropriate for this procedure.
20. Subjects that have life expectancy < 90 days, in the opinion of the investigator at the time of enrollment.
21. Subjects dependent on extracorporeal life support such as extracorporeal membrane oxygenation (ECMO).
22. Participation in another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of Device-Related Adverse Events (AEs) | Through 30 days post-procedure
  The number and proportion of subjects who experienced at least one device-related adverse event. This will be summarized, and the 95% confidence interval of the proportion will be presented. The incidence of device-related adverse events by type and seriousness through 30 days will also be summarized.
Rate of Technical Success | Periprocedural
  Successful autologous blood transfusion using the AlphaReturn Blood Management System

SECONDARY OUTCOMES:
Rate of Major Adverse Events (MAEs) | Through 48 hours post-procedure
  The rate of MAEs within the first 48 hours after the index procedure. MAEs include device-related death, major bleeding, and device-related SAEs of clinical deterioration, pulmonary vascular injury, and cardiac injury.
Rate of Complications | Through 48 hours post-procedure
  Rate of complications including device-related clinical deterioration, device-related cardiac injury, device-related pulmonary vascular injury, major bleeding, and device-related death within 48 hours of the index procedure.
Rate of Device-Related SAEs | Through 30 days post-procedure
  Rate of device-related Serious Adverse Events (SAEs) and death for any cause within 30 days post procedure.
Rate of Symptomatic PE recurrence within 30 days | Through 30 days post-procedure
  Symptomatic PE recurrence within 30 days.
Reduction in RV/LV Ratio | Through 48 hours post-procedure
  Reduction in RV/LV ratio between baseline and 48 hours post procedure assessed by CTA.
Thrombolytics Use | Through 48 hours post-procedure
  Use of thrombolytics during or within 48 hours of the procedure.
Length of Stay in Intensive Care Unit | Through 30 days post-procedure
  Length of stay in the Intensive Care Unit (ICU) within 30 days post-procedure.
Length of Stay in Hospital | Through 30 days post-procedure
  Length of stay in the hospital within 30 days post-procedure.